CLINICAL TRIAL: NCT00897169
Title: A Trial Investigating the Possible Difference in the Development of Type 2 Diabetes in Caucasian and Japanese Subjects by a Model-based Analysis
Brief Title: A Trial Investigating the Possible Difference in Development of Type 2 Diabetes Between Caucasian and Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS-3662
Record Dates: First submitted 2009-02-24; First posted 2009-05-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Other: Oral Glucose Tolerance Test (OGTT)
- B (Experimental)
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Other: Euglycaemic hyperinsulinaemic clamp

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — A 5-hour oral glucose tolerance test (OGTT) is performed at visit 2
Other: Euglycaemic hyperinsulinaemic clamp — A 4-hour euglycaemic, hyperinsulinaemic clamp is performed at visit 3
  Arms: B

SUMMARY:
This trial is conducted in Europe and Japan. The aim of this clinical trial is to investigate the possible difference in the development of type 2 diabetes in a Japanese and a Caucasian population. Healthy subjects, subjects with impaired glucose tolerance, as well as subjects with type 2 diabetes will be included in the trial. The development of type 2 diabetes across the cohort will be investigated with regard to insulin sensitivity and B-cell capacity.

ELIGIBILITY:
Inclusion Criteria:

* Danish (Northern European) or Japanese (according to country allocation) background for at least 3 generations
* BMI above or equal to 18 kg/m2

Exclusion Criteria:

* Treatment of diabetes mellitus with any insulin product
* Fasting plasma/serum glucose above 12 mM
* Therapy with TZD (thiazolidinedione) drugs within the past 3 months
* Therapy with more than 2 OADs (oral anti-diabetics drugs)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Beta-cell function index estimated by a model-based analysis fit to the complete OGTT C-peptide and glucose profiles (12 time points), and including diabetes progression (as assessed by the glucose concentration 2 hours after an oral glucose load) | At 5-hour Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Insulin sensitivity estimated by a model-based analysis fit to the complete OGTT insulin and glucose profiles (12 time points) | At 5-hour OGTT and 4-hour clamp procedure
Fraction of the possible difference in ß-cell function and insulin sensitivity between Japanese and Caucasian that can be explained by each covariate factor | At 5-hour OGTT and 4-hour clamp procedure
Evaluation of comparability of OGTT and clamp data based on modelling data of insulin sensitivity from steady-state clamp insulin and glucose concentrations and OGTT insulin and glucose profiles (12 time points) | At 5-hour OGTT and 4-hour clamp procedure

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, København Ø, Denmark
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Moller JB, Pedersen M, Tanaka H, Ohsugi M, Overgaard RV, Lynge J, Almind K, Vasconcelos NM, Poulsen P, Keller C, Ueki K, Ingwersen SH, Pedersen BK, Kadowaki T. Body composition is the main determinant for the difference in type 2 diabetes pathophysiology between Japanese and Caucasians. Diabetes Care. 2014;37(3):796-804. doi: 10.2337/dc13-0598. Epub 2013 Oct 15. PMID 24130359
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com